CLINICAL TRIAL: NCT00275483
Title: Prevention of PONV by Acupressure. A Study of the Effect of a Recently Generated Danish Bracelet Vital-Band(R) Which Stimulates the Acupressure Point P6
Brief Title: Prevention of Postoperative Nausea and Vomiting (PONV) by Acupressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Vital-band 01
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Postoperative Nausea and Vomiting; Acupressure Point P6
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

INTERVENTIONS:
Device: Vital-band (R)

SUMMARY:
The purpose of this study is to determine whether stimulation to the akupressurpoint P6 with a recently developed bracelet are effective preventing postoperative nausea and vomiting

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Non-smoker,
* >18 years,
* ASA 1 or 2,
* Signed patient information,
* IV-anaestesia.

Exclusion Criteria:

* Male,
* Smoker,
* ASA 3 or 4,
* Pregnancy,
* Nausea and vomiting within the last 24 h before operation,
* Diabetes,
* Carpaltunnel syndrome,
* Lymphedema of arms,
* Eczema of forearm,
* Patients who earlier has undergone removal of lymph nodes in the armpits,
* Inhalation anaestesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-05; Primary Completion 2005-10 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting

SECONDARY OUTCOMES:
1: The use of conventionel antiemetic treatment.
2: Lenght of stay in the perioperative unit.
3: overall lenght of stay

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Majholm, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev University Hospital, department of anaestesiology, Copenhagen, Herlev, Denmark